CLINICAL TRIAL: NCT02818816
Title: A Prospective Study to Evaluate the Effect of Preoperative Topical Brimonidine Tartrate 0.2% (Allergan, Irvine, CA) on Intraocular Pressure (IOP) of Patients Undergoing Robot-assisted Laparoscopic Prostatectomy (RALP)
Brief Title: Preoperative Brimonidine on IOP of Patients Undergoing RALP
Acronym: IOPsTBURG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-9684
Record Dates: First submitted 2016-06-22; First posted 2016-06-30 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Prostate Cancer
Keywords: Brimonidine tartrate; Intraocular pressure; Prostate Cancer; Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brimonidine Tartrate; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brimonidine Tartrate 0.2% (2mg/mL) (Experimental): One (I) drop of brimonidine tartrate 0.2% (2mg/mL) will be placed in the randomized eye preoperatively thirty minutes before robotic-assisted radical laparoscopic prostatectomy (RALP)
  Interventions: Drug: brimonidine tartrate 0.2%
- Carboxymethylcellulose Eye Drops (Placebo Comparator): One drop of Carboxymethylcellulose eye drops will be placed in the randomized eye half an hour before RALP
  Interventions: Other: Carboxymethylcellulose Eye Drops

INTERVENTIONS:
Drug: brimonidine tartrate 0.2% — Alpha adrenergic receptor agonist
  Other Names: Alphagan, Allergan, Irvine, CA
  Arms: Brimonidine Tartrate 0.2% (2mg/mL)
Other: Carboxymethylcellulose Eye Drops — Ocular lubricants
  Other Names: Refresh Optive Fusion; Tear drops
  Arms: Carboxymethylcellulose Eye Drops

SUMMARY:
Patients with prostate cancer undergoing robot assisted radical laparoscopic prostatectomy (RALP) in steep Trendelenburg position (sTBURG) are noted to have elevated intraocular pressures (IOP) intraoperatively. One study showed an increase in IOP of 13 millimeters of mercury (mmHg) from baseline IOP levels intraoperatively. Other studies have shown the IOP to more than double intraoperatively during RALP in sTBURG. IOP is found to be directly related to angle of inclination and increases time dependently with sTBURG. The IOP may remain significantly elevated until the first postoperative day after RALP.

There are no previously published data concerning the safe threshold for IOP elevation and the effects of this increased IOP on vision and on generalized eye health are still not entirely known. One study showed postoperative visual field defects in 28% (7/25) of patients who underwent RALP in sTBURG. It has been theorized that sTBURG and subsequent increased IOP are risk factors for postoperative vision loss (PVL). It is believed that the increased IOP decreases optic nerve perfusion pressure causing ischemic optic neuropathy. Some previously recommended ways to reduce the intraoperative IOP spike during RALP include shorter operating times, decreased angle of inclination, modified Trendelenburg position, use of Propofol for maintenance anaesthesia and intraoperative topical hypotensive agents to reduce IOP. Given the challenges with some of the above options, this study aims to evaluate the effect of pre-operative treatment with topical Brimonidine Tartrate 0.2% on the IOP of patients undergoing RALP with sTBURG. The goal is to prevent the anticipated IOP spike thereby reducing risk of postoperative vision loss.

DETAILED DESCRIPTION:
With completed informed consent, study participants will undergo a pre-operative comprehensive ophthalmic evaluation to document best corrected visual acuity (VA), IOP measurements, visual field assessments (VF), optical coherence tomography measurements (OCT) of the retinal nerve fiber layer, optic disc photography and screening for other ophthalmologic abnormalities. Height and weight measurements will also be recorded.

Using opaque envelopes with the aid of Sequentially Numbered Opaque Sealed Envelopes (SNOSE) schemes, each patient will be randomized to either right eye or left eye. Thereafter patients will be randomized to placebo (carboxymethylcellulose) or drop (Brimonidine tartrate 0.2%) which will be given 30 minutes before the start of surgery with the patient in horizontal supine position. Eyes randomized to receive a drop will be treated with one drop of Brimonidine tartrate 0.2% while eyes randomized to receive placebo will receive one drop of Carboxymethylcellulose eye drops (Control group).

IOP measurements will be recorded for both eyes pre-operatively in the upright seated position (baseline), pre-anaesthetized in supine horizontal position, intra-operatively in anaesthetized supine horizontal position, hourly intra-operatively in anaesthetized sTBURG, awake post-operatively in supine horizontal position and at 1 month postoperatively in the upright seated position. Three IOP measurements will be recorded, each with 5% confidence interval (CI). Blood pressure and end tidal carbon dioxide will be recorded hourly intra-operatively. The following surgical data will also be recorded: procedure duration, angle of inclination of surgical bed, anesthetic agents used, fluid volume given, transfusions given, blood loss volume and complications. Best corrected VA, IOP, VF, OCT and optic disc photography will also be recorded for each patient at the 1-month post-operative visit.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18 years and above
* Patients with a diagnosis of prostatic carcinoma requiring prostate surgery

Exclusion Criteria:

* Patients having had an ophthalmic surgical procedure within 6 months of the beginning of the study.
* Patients with a diagnosis of glaucoma
* Any abnormality of the cornea which may prevent reliable applanation tonometry
* Known allergy/ hypersensitivity reaction to Brimonidine
* Contra-indication to Brimonidine including patients on monoamine oxidase inhibitors (MOA)
* Patients unwilling or unable to provide informed consent
* Patients with anticipated difficult airway management (as this may require medications and/or airway manipulations resulting in increased IOP)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2017-01-24 (Actual); Study Completion 2017-08-07 (Actual)

PRIMARY OUTCOMES:
Changes in IOP during the course of the surgical procedure between eyes treated with medication and those with placebo with patients undergoing RALP with sTBURG | Preoperatively within 1-2 months, intraoperatively, and postoperatively within 1-2 months
  Changes in IOP during the course of the surgical procedure between eyes treated with medication and those with placebo with patients undergoing RALP with sTBURG

SECONDARY OUTCOMES:
Changes in Visual acuity, visual fields, retinal nerve fiber layer thickness | Preoperatively within 1-2 months, intraoperatively, and postoperatively within 1-2 months
  Changes in Visual acuity, visual fields, retinal nerve fiber layer thickness when preoperative and postopertive evaluations are compared

CONTACTS AND LOCATIONS:
Overall Officials: Buys M Yvonne, MD FRCSC, Principal Investigator — University of Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No